CLINICAL TRIAL: NCT00821743
Title: Study of Deep Brain Stimulation of the Pedunculo-pontin Nucleus (PPN) for the Treatment of Gait and Balance Disturbances in Patients With Parkinson's Disease (PPN-GAB-PARK Study)
Brief Title: Pedunculo-Pontin Nucleus (PPN) - Deep Brain Stimulation (DBS) in Gait and Balance Disturbance in Parkinson's Disease (PPN-GAB-PARK Study)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PPN-GAB-PARK study
Record Dates: First submitted 2009-01-12; First posted 2009-01-13 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2010-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): The DBS electrodes (model 3389, Medtronic) will be stereotactically implanted bilaterally in the PPN, according to the technique usually used for STN-DBS, and connected to the subcutaneously implanted stimulator (Kinetra, Medtronic).
  Interventions: Device: Deep brain stimulation electrode

INTERVENTIONS:
Device: Deep brain stimulation electrode — The DBS electrodes (model 3389, Medtronic) will be stereotactically implanted bilaterally in the PPN, according to the technique usually used for STN-DBS, and connected to the subcutaneously implanted stimulator (Kinetra, Medtronic).

SUMMARY:
Disturbance of posture, gait and balance usually appear several years after Parkinson's disease (PD) onset. These axial signs, generally resistant to conventional drug and non-drug treatment, can generate a loss of autonomy and traumatic complications. Improvement of these axial signs by deep brain stimulation (DBS) of the pedunculo-pontin nucleus (PPN) has been described for a small number of patients. The objectives of the present prospective monocentric pilot study are to determine the optimal stimulation parameters of PPN-DBS, to evaluate the long term tolerance and the effect of PPN-DBS on axial signs and quality of life in five patients with severe PD. The use of detailed clinical rating scales and quantitative computer-based gait analysis will allow to identify the optimal stimulation parameters and relevant clinical efficacy parameters, mandatory for the design of further comparative large-scale studies.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a neurodegenerative disorder with an association of akinesia, rigidity and tremor, but also so-called "axial" motor signs (disturbance of posture, gait and balance) that usually appear after several years of disease evolution. These axial signs, generally resistant to drug treatment and deep brain stimulation (DBS) of subthalamic nucleus (STN), can generate a loss of autonomy and traumatic complications due to frequent falls. An improvement of axial signs by DBS of the pedunculo-pontin nucleus (PPN) has been described for a small number of patients. Nevertheless, this effect needs to be confirmed in more patients and there is need for complementary knowledge, including optimal stimulation modalities.

The primary objective of the current prospective monocentric pilot study is to determine the optimal stimulation parameters (site of stimulation, frequency, amplitude) of PPN-DBS in patients with severe PD. Secondary objectives are 1) to confirm the effect of PPN-DBS on disturbance of posture, balance and gait; 2) to evaluate long term tolerance of this technique; 3) to determine the components of gait that are most improved by PPN-DBS; 4) to evaluate unilateral versus bilateral stimulation; 5) to evaluate the effects of PPN-DBS on other PD symptoms; 6) to determine the impact of PPN-DBS on quality of life. Five patients fulfilling the following criteria, will be included: age between 18 and 70 years, idiopathic PD for more than 5 years, predominant axial motor signs (disturbance of gait and balance, falls, freezing of gait) responsible for disability in daily living and resistant to optimal treatment.

The DBS electrodes (model 3389, Medtronic) will be stereotactically implanted bilaterally in the PPN, according to the technique usually used for STN-DBS, and connected to the subcutaneously implanted stimulator (Kinetra, Medtronic). After the surgery, the study will comprise two phases: a 6-month phase dedicated to optimisation of the stimulation parameters (including systematic evaluation of defined parameters); followed by a phase of evaluation, that will compare, in a double-blind setting, 4 conditions (right unilateral, left unilateral, bilateral and off stimulation). Efficacy of PPN-DBS will be evaluated by clinical rating scales quantifying motor disturbance, cognitive function and quality of life, and by the means of computer-based measure of gait and balance (system Gaitrite and Vicon).

Expected results are 1) an improvement of gait, postural and balance disturbance, due to PPN-DBS. 2) Identification of the optimal PPN-DBS parameters, improving most the axial PD symptoms, will allow to abbreviate the adjustment period, by using as default setting these parameters when turning on the stimulator for the first time; 3) Identification of the axial signs which are the most improved will allow to select patients that could most benefit from PPN-DBS 4) The use of diverse specific rating scales and quantitative gait analysis will allow to determine the most relevant clinical criteria to be evaluated in further studies.

Thus, this project will allow to obtain data (selection criteria, relevant rating scales, optimal stimulation parameters) mandatory for the construction of further comparative large-scale studies, if the efficacy of PPN-DBS was confirmed by the present study.

ELIGIBILITY:
Inclusion Criteria:

* Severe idiopathic Parkinson's disease (stage of Hoehn and Yahr ≥ 3).
* Disease duration ≥ 5 years.
* Predominant axial motor signs (gait and balance disturbance as freezing of gait, postural instability, falls) with disability in daily life, defined by a score UPDRS II 2 of item 13 or 3 of item 14 or 15.
* Axial motor signs resistant to optimal drug and non-drug treatment, including physical therapy and eventually STN-DBS (if STN-DBS is ongoing for at least 1 year and has shown no efficacy on axial motor signs).
* No significant abnormality on brain MRI.

Non-inclusion criteria

* Patient with non-axial, dopa-responsive motor signs and indication of first line STN-DBS. In case of absence of efficacy of STN-DBS on axial motor signs after one year of stimulation, PPN-DBS may be proposed to these patients.
* Patient with major cognitive disturbances defined by a score Mattis DRS 130 (of 144).
* Pregnant or breast-feeding woman.
* Patient with contraindication for general anaesthesia, a contraindication for surgery (including disorders of haemostasis, or necessity of anticoagulant and antiaggregant drug), or a contraindication for MRI.
* Patient presenting major depression, psychosis or addiction in six months preceding inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2010-03; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint will be the optimal parameters of PPN-DBS, defined as those leading to the best improvement of posture, balance and gait disturbance | at day 0, day 7, 6 months, year 1 and year 2

SECONDARY OUTCOMES:
Efficacy of PPN-DBS on disturbance of posture, balance and gait | at day 0, day 7, 6 months, year 1 and year 2
Long term tolerance will be assessed by general and neurological examination, neuro-psychological tests (MMS, Mattis-DRS, Score fontal, BREF, MADRS) and by assessment of adverse events; | at day 0, day 7, 6 months, year 1 and year 2
the components of gait that are most improved by PPN-DBS will be determined using computer-based systems (GAITRite and VICON); | at day 0, day 7, 6 months, year 1 and year 2
evaluation of unilateral versus bilateral stimulation will be done during the double-blind assessment of all efficacy criteria; | at day 0, day 7, 6 months, year 1 and year 2
effects of PPN-DBS on other PD symptom will be assessed using UPDRS and Hoehn and Yahr's staging; | at day 0, day 7, 6 months, year 1 and year 2
the impact of PPN-DBS on quality of life and activities of daily living will be assessed by UPDRS II, SF36 and PDQ39 questionnaires and by a global satisfaction scale. | at day 0, day 7, 6 months, year 1 and year 2

CONTACTS AND LOCATIONS:
Overall Officials: Denys FONTAINE, PhD, Principal Investigator — Department of neurosurgery, CHU de Nice
Locations (1):
- Neurology, Neurosugery of Nice University Hospital, Nice, France